CLINICAL TRIAL: NCT07236242
Title: Impact of Mothers Consuming a Fennel Infusion on Infantile Colic in Exclusively Breastfed Infants
Brief Title: Effect of Breastfeeding Mothers Drinking Fennel Seed Infusion on Infants With Colic
Acronym: BabyGut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IITAA, Universidade dos Açores (Other)
Responsible Party: Principal Investigator, Celia Costa Silva, Professor, IITAA, Universidade dos Açores
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M1.1.C/C.S./050/2021/01
Record Dates: First submitted 2025-09-26; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Colic, Infantile
Keywords: Fennel
MeSH Terms: conditions — Colic

STUDY DESIGN:
Masking Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mother - Infant (Experimental): Breastfeeding women and their infants
  Interventions: Dietary Supplement: Fennel infusion

INTERVENTIONS:
Dietary Supplement: Fennel infusion — The mothers were asked to drink an infusion of fennel seeds (1 L per day) for one week .

SUMMARY:
The goal of this clinical trial is to determine whether a fennel-water infusion taken by mothers reduces colic in breastfed infants. The study will also assess the effect of the fennel infusion on the mothers' milk and the gut microbiota of the infants. The main questions it aims to answer are:

* Does a fennel-water infusion taken by mothers reduce colic in breastfed infants?
* What changes occur in the gut microbiota of responders (participants whose infants show reduced colic symptoms after the intervention)? Researchers will evaluate changes in the microbiota of breast milk and the stool of breastfed infants after the mothers consume a fennel infusion.

Participants-mothers of infants-will:

* Take 1 L of fennel infusion daily for 7 days.
* Keep a diary of infant colic symptoms, including time spent crying, and periods of fussiness or irritability without a definite explanation.
* Provide breast milk and infant stool samples before treatment (day 0) and at the end of treatment (day 7) for analysis of microbial communities.

DETAILED DESCRIPTION:
The project will investigate the effect of maternal ingestion of fennel infusion and the associated microbial changes in milk and the infant gut. A beneficial effect has been reported by mothers as part of popular medicine, but this has not been studied in controlled trials.

The trial aims to elucidate the mechanisms by which fennel compounds exert a colic-reducing effect in babies via breast milk. The investigators will determine whether an orally administered fennel seed infusion affects monitored symptoms or microbial parameters, and whether the composition of the fecal microbiota differs between colicky and non-colicky infants. Mothers will be asked to drink an infusion of fennel seeds (Foeniculum vulgare var. dulce) (20 g/L, 1 L per day) for one week. Samples of milk and feces will be collected at the beginning of treatment (day 0) and at the end of treatment (day 7) for microbiome analysis.

Samples will be prepared for Illumina sequencing by 16S rRNA gene amplification of the bacterial community. Raw reads will be extracted from the Illumina MiSeq System in fastq format and processed in the QIIME2 package using DADA2 to infer amplicon sequence variants (ASVs) and their relative abundances across samples. Taxonomy will be assigned to ASVs with the q2 feature-classifier using a pre-trained Naïve Bayes classifier of the Silva database. For species assignment, sequences will be further analyzed using the GenBank DNA database with the Basic Local Alignment Search Tool (BLAST) algorithm.

Alpha diversity will be determined using the number of taxa, individuals - amplicon sequence variants (ASVs), dominance (1-Simpson index), Margalef's richness index, evenness, and Chao1. Alpha diversity results will be compared before and after the intervention using the Wilcoxon signed-rank test. Beta diversity will be measured using principal coordinate analysis (PCoA) based on Bray-Curtis distance matrices for ASVs and PERMANOVA. The Wilcoxon signed-rank test will be used to compare normalized ASVs at the genus and species levels before the intervention (day 0) and after (day 7).

ELIGIBILITY:
Inclusion Criteria:

* Breastfed infants aged 1 to 5 months, full-term (gestational age between 38 and 42 weeks) of both sexes, diagnosed with infantile colic. The ROME IV criteria for diagnosed infant colic were used in this study.

Exclusion Criteria:

* Infants fed with artificial infant formula, use of antibiotics in the last 3 months by mothers or infants.

Ages: 1 Month to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a ≥50% reduction in daily crying duration as measured by a parent-reported 24-hour diary. | One week
  Response is defined as a reduction of at least 50% from baseline in mean daily crying duration. The baseline value is the mean daily crying duration recorded by parents in a 24-hour diary for the two days before treatment initiation, as reported in a questionnaire. The post-treatment value is the mean daily crying duration recorded in the 24-hour diary on the final two days of the one-week treatment period.
Changes in bacterial community of infant stool samples | One week
  The bacterial community, assessed by changes in biodiversity indices and the relative proportions of bacterial genera in infant stool samples, will be evaluated before the intervention (day 0) and at the end of the trial (day 7).

SECONDARY OUTCOMES:
Changes in bacterial community of breast milk | One week
  The bacterial community, assessed by changes in biodiversity indices and the relative proportions of bacterial genera in breast milk samples, will be evaluated before the intervention (day 0) and at the end of the trial (day 7).

CONTACTS AND LOCATIONS:
Overall Officials: Célia C. Silva, Principal Investigator — IITAA, Universidade dos Açores
Locations (2):
- Portugal (2):
  - Universidade dos Açores, IITAA, Angra do Heroísmo, Azores
  - Universidade dos Açores, FCAA, Angra do Heroísmo

IPD SHARING:
Plan to Share IPD: No
IPD used in the results publication.

DOCUMENTS (1):
  • Informed Consent Form (2021-04-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT07236242/ICF_000.pdf